CLINICAL TRIAL: NCT00936923
Title: Effect of Diuretics on Fluid Status Control and Residual Renal Function in Peritoneal Dialysis Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn prior to enrollment of first participant.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGPD-diuretics
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Renal Function Disorder
Keywords: CAPD; Diuretics; Residual Renal Function; furosemide
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- furosemide1 (Active Comparator): Patients will take furosemide 60mg per day for 1 years and undergo a study assessment at 3, 6, 12, 18, 24 months .
  Interventions: Drug: furosemide
- furosemide 2 (Active Comparator): Patients will take 120mg furosemide per day for 1 years and undergo a study assessment at 3, 6, 12, 18, 24 months .
  Interventions: Drug: furosemide
- control (No Intervention): Patients in control group will not take furosemide

INTERVENTIONS:
Drug: furosemide — patients will take furosemide 60 or 120mg oral per day for 1 years .
  Other Names: Lasix(Diuretics)
  Arms: furosemide 2; furosemide1

SUMMARY:
A prospective, randomized, open-label, stratified, controlled clinical trial to evaluate whether long term furosemide therapy (1 year) would preserve urine volume and/or residual renal function (RRF) and improve fluid state in continuous ambulatory peritoneal dialysis (CAPD) patients.

DETAILED DESCRIPTION:
There are 3 phases in this study. Phase 1 is screening phase. Each subject will be evaluated to determine if he/she is eligible for the study. Phase 2 is the intervention phage. Patients are divided arbitrarily into two groups according to baseline RRF (residual glomerular filtration rate [rGFR] <5or > 5 ml/min), then randomly received 12 months treatment with the study drugs( furosemide 120mg daily, 60mg daily, or no diuretic). Phase 3 is following-up phase, which lasts 1 year. Dialytic prescription is adjusted independent of the study and is guided by clinical parameters and calculated clearances (target creatinine clearance 65L/week, urea clearance Kt/V > 1.7 per week). Blood pressure is measured using an automated blood pressure device, and the target level is 135/85mmHg. The antihypertensive medication is introduced after the body weigh reduced into target level, and the ACEI and /or ARB selection is needed to the cross-sectional design. The hydration state is measured by bioelectrical impedance analysis (BIA).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Age:20~70 years, regardless of gender
* All patients received CAPD more than 1 months;
* Urine volume of 500ml/d or more;
* No history of taking furosemide for at least 2 weeks .

Exclusion Criteria:

* Inability or unwillingness to sign the informed consent
* Inability or unwillingness to meet the scheme demands raised by the investigators
* Current acute infection such as peritonitis ;
* Severe diarrhea or vomiting within the preceding 1 month
* Acute Cardiac failure
* Myocardial infarction within the preceding 6 months;
* Hypertensive encephalopathy or cerebrovascular accident;
* Accident within the preceding 6 months;
* Any condition, such as alcohol or drug abuse, chronic liver disease, malignant disease, or psychiatric disorder;
* Allergy or intolerance to furosemide .
* Current or recent (within 2 weeks) exposure to any other investigational drugs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Residual renal function and urine volume | Every 3 months

SECONDARY OUTCOMES:
Dialysis adequacy, fluid status(BIA parameters: Total body water, ECW/TBW), serum Cystatin C, blood pressure, hospitalization, death from any cause,cardiovascular events, any adverse drug effects | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD,PhD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China